CLINICAL TRIAL: NCT05922826
Title: Clinical Empirical Research of ARDS
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Chinese PLA General Hospital, Chinese PLA General Hospital
Other Study IDs: ARDS Research
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Invasive Mechanical Ventilation ARDS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to the ARDS Berlin definition, patients with severe concurrent invasive mechanical ventilation were selected, and clinical data and prognosis were collected. Samples such as blood and balf were collected for analysis based on changes in the condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the Berlin definition of ARDS and require invasive mechanical ventilation. ARDS diagnostic criteria: according to the Berlin definition, Chest radiograph shows patchy shadows in the lungs; Respiratory failure cannot be completely caused by heart failure or excessive fluid infusion
2. ARDS onset ≤ 3 days when included in the study
3. Patient PaO2/FiO2 ≤ 200mmHg when included in the study

Exclusion Criteria:

* 1) Patients with intracranial hypertension, pleural fistula, pneumothorax, HIV, HBV, HCV

  2) Age>85 years old or<18 years old

  3) Pregnant patients

  4) Severe hemodynamic instability (vasopressor increase>30% in the first 6 hours, or Norepinephrine>0.5 mg kg/min)

  5) Patients unable to perform EIT ventilation and/or perfusion testing (unable to perform internal jugular vein catheterization, Hypernatremia, chest malformation, active implant device, unstable spinal injury or fracture, skin lesions opposite the EIT monitoring area)

  6) Patients with abnormal esophageal anatomical structure and inability to indwelling gastric tubes

  7) Disagreement for inclusion in this study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the ARDS Berlin definition, patients with severe concurrent invasive mechanical ventilation were selected, and clinical data and prognosis were collected. Samples such as blood and balf were collected for analysis based on changes in the condition.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-18 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary and Critical Care Medicine, Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duan Z, Lian D, Wang K, Hu Y, Fu H, Wen R, Zhao Y, Hu X, Pan P, Xu J, Chen J, Xiao L, Wang L, Yu X, Han X, Xie W, Xie F, Xie L, Han Z. Multi-modal data to identify key factors influencing lung injury in ARDS patients undergoing invasive mechanical ventilation: A prospective multi-center observational study protocol. PLoS One. 2026 Jan 23;21(1):e0332985. doi: 10.1371/journal.pone.0332985. eCollection 2026. PMID 41575959